CLINICAL TRIAL: NCT00594633
Title: Adjunctive Donepezil Therapy and Genetic Risk Factors of Cognitive Dysfunction in Brain Tumor Survivors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-122
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Brain Tumor; Brain Cancer; Cns Cancer; Cognitive Dysfunction
Keywords: Cognitive dysfunction
MeSH Terms: conditions — Brain Neoplasms; Central Nervous System Neoplasms; Cognitive Dysfunction | interventions — Donepezil

ARMS (1):
- 1 (Experimental): donepezil and questionaires
  Interventions: Other: donepezil and questionaires

INTERVENTIONS:
Other: donepezil and questionaires — Patients will undergo a brief cognitive evaluation prior to (baseline/Time 1), Cognitive Re-Evaluation (about 12 weeks after Time 1), Cognitive Re-Evaluation (about 12 weeks after Time 2) ,Cognitive Re-Evaluation (about 6 months after discontinuation of Donepezil). Then pt will be tx with donepezil, an acetylcholinesterase inhibitor. They will undergo a four-week dose titration (i.e., 5mg QD during weeks 1-4) to reach a final dose of 10mg QD of oral donepezil there after for a maximum of 24 weeks.

SUMMARY:
A significant number of brain tumor patients who received radiation or chemotherapy have thinking problems as a result of their treatment. The purpose of this study is to find out if treatment with Aricept (donepezil) may improve some aspects of thinking abilities in patients with brain tumors who received radiation or chemotherapy. This research will also study whether persons having particular genes for a blood-borne substance called apolipoprotein E (APOE) are more likely to have thinking problems after radiation or chemotherapy treatment for their brain tumors. The findings of this study will help us find out whether Aricept can improve thinking abilities after cancer treatment, and whether some of the thinking difficulties may be in part related to having certain genes.

DETAILED DESCRIPTION:
A significant proportion of brain tumor patients treated with radiation or chemotherapy who are in disease remission experience cognitive sequelae from their treatment. Cognitive dysfunction can be of sufficient severity to interfere with their ability to function at premorbid professional and social levels. There are, however, no approved pharmacological interventions for improving cognitive functions in cancer patients who display treatment-related cognitive deficits. Donepezil, an acetylcholinesterase inhibitor, has been shown to provide cognitive and functional benefits in patients with Alzheimer's disease, vascular dementia, and in patients with other neurological diseases without known cholinergic deficiency. The proposed pilot study will examine the efficacy of donepezil in improving cognitive functions in adult brain tumor patients treated with radiation and/or chemotherapy who have mild to moderate cognitive difficulties. Neuropsychological measures of executive, psychomotor speed, attention, and memory abilities will be administered prior to, during and following donepezil therapy. The proposed study will also test the hypothesis that the apolipoprotein E (APOE) e-4 allele correlates with the development of cognitive impairment after radiation or chemotherapy treatments. The proposed investigation is unprecedented and may provide preliminary information about (1) a pharmacological therapy that could improve cognitive functions in this population, and (2) a genetic risk factor that may increase vulnerability to radiation or chemotherapy-induced cognitive decline.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with a brain tumor and treated with cranial irradiation and/or chemotherapy, and in stable remission of their disease at the time of enrollment.
* completed radiation and/or chemotherapy treatment at least 6 months prior to being enrolled in the study.
* who obtain a Mini-Mental Status Examination (MMSE) score ranging from 18 to 28 at the time of enrollment.
* are at least 18 years of age.
* are English speaking.
* have capacity to give consent

Exclusion Criteria:

* Patients with active or progressive disease on recent MRI of the brain either at the time of enrollment, or during the study period.
* with a pre-existing uncontrolled seizure disorder, or significant renal or hepatic impairment.
* taking the following medications: antipsychotics, psychostimulants.
* patients who have been on selective serotonin re-uptake inhibitors (SSRIs) for less than 3 months at the time of enrollment.
* with uncontrolled behavioral or mood disturbances.
* have their anticonvulsant medication(s) or dosage(s) changed less than 30 days prior to enrollment.
* currently receiving donepezil or other cholinesterase inhibitors.
* who is pregnant.
* unable to cooperate or complete cognitive tests.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2004-10; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
The primary goal of this study is to assess the efficacy of donepezil in improving executive abilities and psychomotor speed in adult brain tumor patients who have undergone cranial irradiation and/or chemotherapy. | conclusion of study

SECONDARY OUTCOMES:
This study will also assess the efficacy of donepezil in improving other cognitive domains such as attention, memory, and general cognition in this population. | conclusion of study
The study will also explore the possibility that the possession of the apolipoprotein E (APOE) є-4 allele is associated with the development of cognitive difficulties following cranial radiation and/or chemotherapy treatments. | conclusion of study

CONTACTS AND LOCATIONS:
Overall Officials: Denise Correa, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org